CLINICAL TRIAL: NCT04762342
Title: Power Training in Older Multiple Sclerosis Patients
Acronym: POTOMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University of Southern Denmark (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4168624
Record Dates: First submitted 2021-02-05; First posted 2021-02-21 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis; Sclerosis; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Demyelinating Diseases; Healthy Aging; Aging
Keywords: Multiple Sclerosis; Healthy aging; Exercise; Neuroprotection
MeSH Terms: conditions — Multiple Sclerosis; Sclerosis; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Demyelinating Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group Multiple Sclerosis (Experimental): 24 weeks of moderate to high-intensity power training (resistance training- emphasizing an explosive concentric phase of muscle contraction) performed twice weekly.
  Balance- and functional exercises are included after week 8.
  Interventions: Other: Power training
- Control Group Multiple Sclerosis (No Intervention): Habitual lifestyle including standard care.

INTERVENTIONS:
Other: Power training — First a brief warm up on a stationary bike and uni-lateral knee raises is completed.
  Power training: Involves exercises performed with fast/explosive muscle contraction during the concentric phase, and slow/controlled (approximately 2-3 s) muscle contraction during the eccentric phase.
  Functional- and balance exercises are included from week 9-24.
  Progression:
  Week 1-4: 3 sets of 12 repetitions at a load of 14 repetitions maximum (RM) with focus on introducing resistance exercise and familiarizing participants with exercises.
  Week 5-8: 3 sets of 12 repetitions at a load of 14 RM the power training component.
  Week 9-16: 3 sets of 10 repetitions at a load of 12 RM. Week 17-24: 3 sets of 8 repetitions at a load of 10 RM
  Strengthening exercises:
  * Bilateral leg-press
  * Bilateral plantar flexion
  * Bilateral knee extension
  * Unilateral banded dorsal flexion
  * Bilateral lying leg curl
  * Back extension
  * Shoulder press
  * Seated row
  * Chest press
  * Lat pull-down
  Arms: Training Group Multiple Sclerosis

SUMMARY:
The study seeks to investigate whether 24 weeks of power training has neuroprotective effects in older PwMS. Additional purposes are to examine the effects of 24 weeks power training on physical function, cognitive function and neuromuscular function. Further, it is investigated whether the potential effects of power training are maintained after 24 weeks of follow-up.

DETAILED DESCRIPTION:
Over the past 3-4 decades, the lifespan among people with multiple sclerosis (MS) has increased substantially. Today more than one-third of all people with MS are 60 years or older. With advanced age, people with MS are more likely to have impairments in cognitive and physical function.

Positive adaptations within the nervous system (~neuroplasticity) have been shown to occur in people with MS following periods of resistance training (RT). This resembles the observations in young and old healthy individuals. Moreover, a specific type of RT termed power training appears to be particularly beneficial, as it emphasizes an explosive concentric phase of muscle contraction. This taxes the nervous system to a very high extent. As a result, power training has been shown to improve several aspects that rely on the nervous system in older individuals without MS. These aspects include cognition, neuromuscular function, and physical function.

The investigators speculate that older people with MS would also benefit. However, no studies have looked into the effects of power training in older people with MS.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 60 years of age.
* Clinically diagnosed with MS according to the McDonald criteria (48).
* Having an EDSS ≤ 6.5.
* able to transport themselves to the testing at Aarhus University and Aarhus University Hospital.
* able to transport themselves to training, if randomized to the PRP group.

Exclusion Criteria:

* having comorbidities (cardiovascular, respiratory, orthopedic, or other neurological diseases than MS) affecting PRP participation or MRI scans.
* having a pacemaker.
* having metallic implant(s) that prevents MRI scans.
* having untreated osteoporosis; t-score below -2.5 and a history of low energy facture or t-score below -3.0.
* participating in more than two sessions per week of structured PRE and have done so for the past 3 months.
* Are cognitively impaired at a level expected to prevent the participant from understanding training and testing instructions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2024-08-28 (Estimated); Study Completion 2024-08-28 (Estimated)

PRIMARY OUTCOMES:
Percentage brain volume change. | Baseline, after 24 weeks and after 48 weeks.
  Whole brain atrophy will be measured from MRI-scans.

OTHER OUTCOMES:
Normalized gray and white matter volume change. | Baseline, after 24 weeks and after 48 weeks.
  MRI scan.
Volume of the brain nucleis: thalamus, hippocampus, putamen, caudate, globus pallidus, corticospinal tract, cingulate gyrus, corpus callosum, cervical spinal volume, motor cortex | Baseline, after 24 weeks and after 48 weeks.
  MRI scan.
Diffusivity of the brain nucleis: thalamus, hippocampus, putamen, caudate, globus pallidus, corticospinal tract, cingulate gyrus, corpus callosum, cervical spinal volume, motor cortex | Baseline, after 24 weeks and after 48 weeks.
  DTI scan.
White matter fibre orientations | Baseline, after 24 weeks and after 48 weeks.
  MKI scan.
Glial fibrillary acidic protein (GFAP) change. | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample- Marker of neurodegeneration.
Neurofilament light chain (NfL) change. | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample-Marker of neurodegeneration:
Brain-derived neurotrophic factor (BDNF) change. | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample-Neurotrophic factor.
Insulin-like growth factor-1 (IGF). | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample-Neurotrophic factor.
C-reactive protein (CRP) change. | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample-Inflammatory markers.
Interleukin-6 (IL-6) change. | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample-Inflammatory markers.
Tumor necrosis alpha (TNF-alpha) change. | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample-Inflammatory markers.
C-terminal collagen cross-links (CTX) change. | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample- Bone turnover markers.
Type-1n-terminal propeptide (P1NP) change. | Baseline, after 24 weeks and after 48 weeks.
  Resting blood sample- Bone turnover markers.
Bone mineral density of the femoral neck and lumbar spine change. | Baseline, after 24 weeks and after 48 weeks.
  Dexa scan.
Body composition change. | Baseline, after 24 weeks and after 48 weeks.
  Dexa scan- whole body scan.
Cognition change . | Baseline, after 24 weeks and after 48 weeks.
  Selective Reminding Test (memory) and Symbol Digit Modalities Test (processing speed).
Nine step stair test change. | Baseline, after 24 weeks and after 48 weeks
  Time to climb a 9 step flight of stairs.
Six Spot Step Test (SSST) change. | Baseline, after 24 weeks and after 48 weeks.
  SSST is a measure of walking ability, balance and coordination. Measured as the time to complete the course.
Six-minute walk test (&MWT) change. | Baseline, after 24 weeks and after 48 weeks.
  Distance covered on a 30 meter track during six minutes maximal walking. Distance covered each minute is noted.
Timed 25-Feet Walk Test (T25FWT) change. | Baseline, after 24 weeks and after 48 weeks.
  Time to walk 25 feet (normal walk and maximal walk pace).
Short Physical performance battery change. | Baseline, after 24 weeks and after 48 weeks.
  Composite score from Five Times Sit- to- Stand Test, Tandem Test and 3 meter walk test.
Maximal Voluntary Contraction (MVC) change. | Baseline, after 24 weeks and after 48 weeks.
  The following muscle groups are tested: Knee flexors, Knee extensors, Plantar flexor and Dorsal flexor.
Rate of force development (RFD) change. | Baseline, after 24 weeks and after 48 weeks.
  The following muscle groups are tested: Knee flexors, Knee extensors, Plantar flexor and Dorsal flexor.
Dynamic Strength change. | Baseline, after 24 weeks and after 48 weeks.
  The following muscle groups are tested: Knee flexors, Knee extensors, Plantar flexor and Dorsal flexor.
Force Steadiness change. | Baseline, after 24 weeks and after 48 weeks.
  Unilateral leg press
Voluntary activation | Baseline, after 24 weeks and after 48 weeks.
  Interpolated twitch technique applied on the quadriceps muscle
Electromyography (EMG) | Baseline, after 24 weeks and after 48 weeks.
  The following muscle groups are tested: Knee flexors, Knee extensors, Plantar flexor and Dorsal flexor.
Grip strength change. | Baseline, after 24 weeks and after 48 weeks.
  Measured by Hand Dynamoter.
SF-12 change. | Baseline, after 24 weeks and after 48 weeks.
  Patient Reported Outcome Measure.
Pittsburg Sleep Qulity Index change. | Baseline, after 24 weeks and after 48 weeks.
  Patient Reported Outcome Measure.
Brief pain inventory change. | Baseline, after 24 weeks and after 48 weeks.
  Patient Reported Outcome Measure.
Baecke Physical Activity change. | Baseline, after 24 weeks and after 48 weeks.
  Patient Reported Outcome Measure.
HADS change. | Baseline, after 24 weeks and after 48 weeks.
  Patient Reported Outcome Measure.
EQ-5D change. | Baseline, after 24 weeks and after 48 weeks.
  Patient Reported Outcome Measure.
FES-I change. | Baseline, after 24 weeks and after 48 weeks.
  Patient Reported Outcome Measure.
Multiple Sclerosis Impact Scale (MSIS-29) change. | Baseline, after 24 weeks and after 48 weeks .
  Patient Reported Outcome Measure (only applicable for people with MS).
Modified Fatigue Impact Scale (MFIS) change. | Baseline, after 24 weeks and after 48 weeks .
  Patient Reported Outcome Measure (only applicable for people with MS).
12-Item MS walking Scale (MSWS-12) change. | Baseline, after 24 weeks and after 48 weeks .
  Patient Reported Outcome Measure (only applicable for people with MS).
Expanded Disability Status Scale (only applicable for people with MS). | Baseline, after 24 weeks and after 48 weeks.
  The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a trained exercise physiologist.
Nine hole peg test | Baseline, after 24 weeks and after 48 weeks.
  Manual dexterity and upper body function
Physical activity | Baseline, after 24 weeks and after 48 weeks.
  Accelerometry (7 days ware time)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Gaemelke, Msc, Principal Investigator — Exercise Biology, Department of Public Health, Aarhus University
Locations (1):
- Tobias Gæmelke, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurwitz BJ. Analysis of current multiple sclerosis registries. Neurology. 2011 Jan 4;76(1 Suppl 1):S7-13. doi: 10.1212/WNL.0b013e31820502f6. PMID 21205683
- [Background] Marrie R, Horwitz R, Cutter G, Tyry T, Campagnolo D, Vollmer T. Comorbidity, socioeconomic status and multiple sclerosis. Mult Scler. 2008 Sep;14(8):1091-8. doi: 10.1177/1352458508092263. PMID 18728060
- [Background] Hvid LG, Strotmeyer ES, Skjodt M, Magnussen LV, Andersen M, Caserotti P. Voluntary muscle activation improves with power training and is associated with changes in gait speed in mobility-limited older adults - A randomized controlled trial. Exp Gerontol. 2016 Jul;80:51-6. doi: 10.1016/j.exger.2016.03.018. Epub 2016 Apr 14. PMID 27090485
- [Background] Aagaard P, Suetta C, Caserotti P, Magnusson SP, Kjaer M. Role of the nervous system in sarcopenia and muscle atrophy with aging: strength training as a countermeasure. Scand J Med Sci Sports. 2010 Feb;20(1):49-64. doi: 10.1111/j.1600-0838.2009.01084.x. PMID 20487503
- [Background] Schoenfeld BJ, Contreras B, Willardson JM, Fontana F, Tiryaki-Sonmez G. Muscle activation during low- versus high-load resistance training in well-trained men. Eur J Appl Physiol. 2014 Dec;114(12):2491-7. doi: 10.1007/s00421-014-2976-9. Epub 2014 Aug 12. PMID 25113097
- [Background] Best JR, Chiu BK, Liang Hsu C, Nagamatsu LS, Liu-Ambrose T. Long-Term Effects of Resistance Exercise Training on Cognition and Brain Volume in Older Women: Results from a Randomized Controlled Trial. J Int Neuropsychol Soc. 2015 Nov;21(10):745-56. doi: 10.1017/S1355617715000673. PMID 26581787
- [Background] Liu-Ambrose T, Nagamatsu LS, Graf P, Beattie BL, Ashe MC, Handy TC. Resistance training and executive functions: a 12-month randomized controlled trial. Arch Intern Med. 2010 Jan 25;170(2):170-8. doi: 10.1001/archinternmed.2009.494. PMID 20101012
- [Background] Reid KF, Martin KI, Doros G, Clark DJ, Hau C, Patten C, Phillips EM, Frontera WR, Fielding RA. Comparative effects of light or heavy resistance power training for improving lower extremity power and physical performance in mobility-limited older adults. J Gerontol A Biol Sci Med Sci. 2015 Mar;70(3):374-80. doi: 10.1093/gerona/glu156. Epub 2014 Sep 8. PMID 25199912
- [Background] Caserotti P, Aagaard P, Larsen JB, Puggaard L. Explosive heavy-resistance training in old and very old adults: changes in rapid muscle force, strength and power. Scand J Med Sci Sports. 2008 Dec;18(6):773-82. doi: 10.1111/j.1600-0838.2007.00732.x. Epub 2008 Jan 30. PMID 18248533
- [Background] Bottaro M, Machado SN, Nogueira W, Scales R, Veloso J. Effect of high versus low-velocity resistance training on muscular fitness and functional performance in older men. Eur J Appl Physiol. 2007 Feb;99(3):257-64. doi: 10.1007/s00421-006-0343-1. Epub 2006 Dec 5. PMID 17146693
- [Background] Earles DR, Judge JO, Gunnarsson OT. Velocity training induces power-specific adaptations in highly functioning older adults. Arch Phys Med Rehabil. 2001 Jul;82(7):872-8. doi: 10.1053/apmr.2001.23838. PMID 11441371
- [Background] Henwood TR, Riek S, Taaffe DR. Strength versus muscle power-specific resistance training in community-dwelling older adults. J Gerontol A Biol Sci Med Sci. 2008 Jan;63(1):83-91. doi: 10.1093/gerona/63.1.83. PMID 18245765
- [Derived] Kupjetz M, Langeskov-Christensen M, Riemenschneider M, Inerle S, Ligges U, Gaemelke T, Patt N, Bansi J, Gonzenbach RR, Reuter M, Rosenberger F, Meyer T, McCann A, Ueland PM, Eskildsen SF, Nygaard MKE, Joisten N, Hvid L, Dalgas U, Zimmer P. Persons With Multiple Sclerosis Reveal Distinct Kynurenine Pathway Metabolite Patterns: A Multinational Cross-Sectional Study. Neurol Neuroimmunol Neuroinflamm. 2025 Nov;12(6):e200461. doi: 10.1212/NXI.0000000000200461. Epub 2025 Sep 18. PMID 40966534
- [Derived] Gaemelke T, Laustsen C, Feys P, Folkestad L, Andersen MS, Jorgensen NR, Jorgensen ML, Jespersen SN, Ringgaard S, Eskildsen SF, Dalgas U, Hvid LG. Effects of power training in older patients with multiple sclerosis on neurodegeneration, neuromuscular function, and physical function. A study protocol for the "power training in older multiple sclerosis patients (PoTOMS) randomized control trial. Contemp Clin Trials Commun. 2024 Feb 19;38:101279. doi: 10.1016/j.conctc.2024.101279. eCollection 2024 Apr. PMID 38444875